CLINICAL TRIAL: NCT04145271
Title: Pre-Hospital Zone 1 Partial Resuscitative Endovascular Balloon Occlusion of the Aorta for Injured Patients With Exsanguinating Sub-diaphragmatic Haemorrhage (P-PRO-Study)
Brief Title: Pre-Hospital Zone 1 Partial Resuscitative Endovascular Balloon Occlusion of the Aorta for Injured Patients With Exsanguinating Sub-diaphragmatic Haemorrhage
Acronym: P-PRO
Status: Completed | Type: Observational
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 271728
Record Dates: First submitted 2019-09-04; First posted 2019-10-30 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Emergencies; Trauma Injury; Trauma, Multiple
MeSH Terms: conditions — Emergencies; Accidental Injuries; Multiple Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Resuscitative Endovascular Balloon Occlusion of the Aorta (REBOA) — Resuscitative Endovascular Balloon Occlusion of the Aorta (REBOA) is a minimally invasive damage control procedure for life-threatening abdominal and/or pelvic haemorrhage. It involves temporary occlusion of the aorta with an endovascular balloon, providing proximal control to the site of vascular injury whilst supporting cerebral and myocardial perfusion

SUMMARY:
It is unknown whether this evolved strategy (Pre-Hospital Zone I P-REBOA) is feasible and with an acceptable safety profile. This study will address this question, therefore informing the design of a prospective multicentre exploratory cohort study followed by a pilot/feasibility multicenter RCT (IDEAL 2B). The IDEAL Framework is an internationally recognised standard, that describes the stages through which interventional therapy innovation normally passes, the characteristics of each stage and the study design types recommended for each

DETAILED DESCRIPTION:
Haemorrhage (bleeding) is the most common cause of preventable death after injury and is responsible for approximately one-third of trauma deaths (of which between 16-29% of such deaths are thought to be preventable).

Resuscitative Endovascular Balloon Occlusion of the Aorta (REBOA) is a minimally invasive damage control procedure for life-threatening abdominal and/or pelvic haemorrhage. It involves temporary occlusion of the aorta with an endovascular balloon, providing proximal control to the site of vascular injury whilst supporting cerebral and myocardial perfusion.

Emergency Department (ED) use of REBOA appears to be feasible and associated with improved outcomes. However, bleeding trauma patients die quickly and it's evident that the peak death rate from haemorrhage occurs within 30 minutes of injury. This is well before the majority of patients can reach hospital, it's therefore likely this resuscitation strategy may have greatest benefit for patients when used in the pre-hospital environment.

We have demonstrated that Pre-Hospital Zone III REBOA (distal aortic occlusion) for exsanguinating pelvic haemorrhage is a feasible resuscitation strategy that significantly improves blood pressure and may reduce the risk of hypovolaemic cardiac arrest and early death due to exsanguination.

To evolve this resuscitation strategy, it is important to establish whether it can be delivered in patients with more proximal haemorrhage in the abdomen (Zone I REBOA). However, this development may be associated with increased risk of harm due to the visceral ischaemia that is created. The use of a technique called Partial REBOA (P-REBOA) may offer a solution by mitigating the ischaemia/reperfusion injury created.

It is unknown whether this evolved strategy (Zone I P-REBOA) is feasible in the pre-hospital setting. This study therefore aims to establish via an Observational Cohort of eight adult trauma patients whether Zone I P-REBOA can be achieved in pre-hospital resuscitation of adult trauma patients with exsanguiunating sub-diaphragmatic haemorrhage at risk of imminent hypovolaemic cardiac arrest or recent hypovolaemic cardiac arrest.

ELIGIBILITY:
Inclusion Criteria -

* Adult trauma patients (aged, or believed to be aged 16 years or older) attended by LAA;
* assessed to have exsanguinating sub-diaphragmatic haemorrhage and imminent risk of hypovolaemic cardiac arrest, or recent hypovolaemic cardiac arrest;
* which is thought to be amenable to treatment with Zone I REBOA;
* and an attempt is made at femoral arterial access (percutaneous access or open surgical approach to insert 8Fr REBOA access sheath)

Exclusion Criteria -

* Age < 16 years
* Injuries deemed clinically unsurvivable
* Known or visible advanced pregnancy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 8 Patients cannulated for REBOA (+ all other patients meeting the inclusion criteria during the study period where there was a failed attempt at femoral arterial access).
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-06-27 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Zone 1 REBOA | 1 day
  The proportion of patients where Pre-Hospital Zone 1 REBOA is achieved, defined as:
  * Balloon insertion depth between 35 - 55 cm
  * Proximal arterial blood pressure transduced
  * Balloon inflation
Partial REBOA (P-REBOA) | 1 day
  The proportion of Pre-Hospital Zone 1 REBOA patients where P-REBOA is achieved, defined as:
  * Evidence of an increase in distal mean arterial pressure (MAP) of at least 5mm - 10mmHg above post inflation baseline;
  * and/or a return of distal pulsatility;
  * or distal pulsatility never absent post initial balloon inflation.

SECONDARY OUTCOMES:
• Incidence of Zone I balloon positioning in the ED | 1 Days
  On routinely performed plain film chest X-Ray. Defined as balloon positioned between T4 - L1 and/or distal to carina, proximal to diaphragm) or on CT.
• Incidence of pre-hospital balloon migration | 1 Day
  (>2cm from the recorded insertion depth, reported by the pre-hospital clinical team
• Incidence of balloon repositioning (proximal or distal) pre or in-hospital. | 1 Day
  Repostioned in aorta for clinical reason
• Method of achieving Partial REBOA | 1 Day
  Balloon deflation, spontaneous, or straight to P-REBOA.
• Incidence of failed femoral arterial access | 1 Day
  Inability to successfully cannulate the CFA percutaneously or via an open approach.
• Time elapsed from balloon inflation to the institution or recognition of P-REBOA. | 1 Day
  Temporal
• Incidence of balloon reinflation or the requirement for additional balloon volume, post institution or recognition of P-REBOA. | 1 Day
  For clinical reason.
• Total duration of REBOA (inflation to final deflation). | 1 Day
  Temporal
• Systolic blood pressure response to institution of REBOA | 1 day
  Physiological
• Incidence of pre-hospital cardiac arrest | 1 day
  Pre and post REBOA, absent carotid or central pulse.
• Incidence of pre-hospital, ED, or operating theatre resuscitative thoracotomy (RT). | 1 Day
  RT
• Mortality rate - Pre-hospital, one hour, 3 hours, 24 hours, 30 and 90 days. | 90 days.
  Mortality
• Causes of death (in-hospital and pre-hospital) of patients who received Pre-Hospital REBOA or did not following a failed attempt. | 1 year
  This will be determined by the SMG following review of all the routinely available clinical information (CT scan results, operative findings and post-mortem findings).
• Survival to hospital discharge. | 90 Days
  Survival
• Length of critical care and hospital stay. | 90 Days
  Temporal
• Incidence of all adverse events related to patient injury, resulting critical illness and treatment as well as femoral cannulation, REBOA catheter insertion and/or the anticipated effects of aortic occlusion: | 90 Days
  * Distal arterial thrombus formation requiring intervention
  * Vascular trauma (related to primary injury or intervention)
  * Surgical repair femoral arterial cannulation site (patch angioplasty)
  * Arterial bypass surgery
  * Cannulation site infection requiring surgical intervention
  * Extremity ischaemia requiring fasciotomies
  * Amputation (primary)
  * Amputation (secondary)
  * Acute renal failure (KDIGO Criteria Stage 3)
  * Requirement for renal replacement therapy (RRT)
  * Acute intestinal ischaemia (Evidence of gut necrosis at laparotomy or findings on CT scanning consistent with gut ischaemia in the context of elevated blood lactate).
  * Multiple Organ Dysfunction Syndrome (MODS, 2 or more organ system failure) including severity of MODS (Sequential Organ Failure Assessment, SOFA Score).

CONTACTS AND LOCATIONS:
Locations (4):
- United Kingdom (4):
  - Royal London Hospital, London
  - London HEMS, London
  - St. Georges Hospital, London
  - St.Marys Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lendrum RA, Perkins Z, Marsden M, Cochran C, Davenport R, Chege F, Fitzpatrick-Swallow V, Greenhalgh R, Wohlgemut JM, Henry CL, Singer B, Grier G, Davies G, Bunker N, Nevin D, Christian M, Campbell MK, Tai N, Johnson A, Jansen JO, Sadek S, Brohi K. Prehospital Partial Resuscitative Endovascular Balloon Occlusion of the Aorta for Exsanguinating Subdiaphragmatic Hemorrhage. JAMA Surg. 2024 Sep 1;159(9):998-1007. doi: 10.1001/jamasurg.2024.2254. PMID 38985496
- [Derived] Lawrie L, Duncan EM, Lendrum R, Lebrec V, Gillies K. Challenges and opportunities for conducting pre-hospital trauma trials: a behavioural investigation. Trials. 2023 Mar 2;24(1):157. doi: 10.1186/s13063-023-07184-5. PMID 36864520